CLINICAL TRIAL: NCT04781283
Title: Prospective Randomized Study Comparing the Kinetics of Endothelial Cell Loss Associated With the XEN® Implant Versus Traditional Filtering Surgery for Glaucoma
Brief Title: Study Comparing the Kinetics of Endothelial Cell Loss Associated With the XEN® Implant Versus Traditional Filtering Surgery for Glaucoma
Acronym: CINEXEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI chose not to start the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CINEXEN
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Glaucoma
Keywords: endothelial cell loss; XEN® implant; filtering surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- specular microscopy (Experimental): The density measurement is a painless and very brief examination (less than a minute) during which the patient places his head on a chin rest while maintaining his forehead on a bar provided for this purpose while looking straight ahead. The measurements are then taken without contact with the patient's eye.
  Interventions: Device: measurement of endothelial cell density by specular microscopy

INTERVENTIONS:
Device: measurement of endothelial cell density by specular microscopy — During this first appointment (T0), in addition to the usual treatment, measurement of the endothelial cell density by specular microscopy will be carried out on the affected eye (basal cell density). To overcome the variability linked to the machine, three consecutive measurements will be taken; the average of the three measurements will be used.
  As part of his post-operative follow-up, the patient will be reviewed at one month, one year, two years, three years, four years and five years after the operation. During these consultations and as part of the research, a new determination of the cell density (3 consecutive measurements) by specular microscopy of the operated eye and an evaluation of the position of the XEN implant will be carried out each time. ® by OCT scan for patients having undergone this surgery.

SUMMARY:
Glaucoma is a blinding optic neuropathy that affects 60 million people worldwide. Of all the types of existing glaucoma, primary open-angle glaucoma is the most common etiology. The therapeutic arsenal today includes drug lowering treatments, lasers and surgery. The most frequent glaucoma surgeries are, in France, trabeculectomy and non-perforating deep sclerectomy (NPDS). These are two filtering surgeries whose principle is to lower the intra ocular pressure (IOP) by creating an evacuation path of the aqueous humor from the anterior chamber (AC) of the eye to the space subconjunctival creating a filtration bubble (FB). These two procedures are currently considered the gold standard. They can be performed alone or at the same time as cataract surgery. The short-term complications encountered with these techniques are early hypotonia and its attendant complications (choroidal detachment, hypotonic maculopathy, hemorrhages, etc.), the most common cause of which is conjunctival leakage from the bubble. In the medium term, increases in blood pressure with deep AC testify to a scleral flap that is too tight which may require suture lysis. Finally, the problems of excessive conjunctival-Tenon healing concern 25 to 30% of those operated on and are responsible for the majority of late blood pressure increases. In the longer term, the most common complication is cataracts; the rarest, but most serious complication is infection of BF, which occurs more readily when the walls of the FB are ischemic or even perforated. It can be complicated by an extremely serious endophthalmitis. A new minimally invasive therapeutic option has been developed limiting per- and post-operative complications. Unlike traditional techniques which present an ab externo approach, the ab interno approach of the new technique proposed consists of the implantation of a tube of collagen 6 mm in length and 45 µm of light called Xen® through the AC .

DETAILED DESCRIPTION:
This surgery can be performed alone or at the same time as cataract surgery. The geometry of the Xen® implant has been studied to help prevent major hypotonia. This new technique would also prevent complications related to conjunctival dissection, while being faster. The placement of a Xen® implant is now used in simple surgery or combined with cataract surgery for open-angle glaucomas, beginners to moderate, associated or not with cataract, progressive and unbalanced under local hypotonizing treatment. Since June 2017, the Xen® technique has been part of the routine in the ophthalmology department of the Paris Saint-Joseph Hospital Group (GhPSJ). The choice of technique (filtering surgery or XEN®) is left to the discretion of the surgeon. To date, no study has yet compared the efficacy and safety of this new technique compared to non-perforating deep sclerectomy: the gold standard. However, the presence of any type of anterior chamber device may be associated with endothelial cell loss even when the device is not in direct contact with the cornea. Endothelial cell loss increases over time well after the operative procedure and sometimes requires removal of the device years later. It can induce non-reversible corneal edema when the device is stopped and involve a corneal transplant. Recently, a study showed that the micro-invasive device ab interno Alcon Cypass® (device similar to XEN®) caused an endothelial cell loss that was not significant initially but significant thereafter (48 months) and not acceptable compared to conventional surgery. glaucoma. The damage was proportional to the area of the implant in the anterior chamber and led to the immediate withdrawal of the device from the market. In view of these results and the absence to date of an equivalent study for XEN®, we proposed to conduct this study in order to assess the possible cell loss compared to NPDS.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥ 18 years
* French-speaking patient
* Patients followed for primary or secondary open-angle glaucoma in the ophthalmology department of the GhPSJ
* Patient with an indication for surgery with placement of Xen® or NDPS alone or combined with cataract surgery by phacoemulsification of the lens
* Patient affiliated to social security or, failing that, to another health insurance system
* Patient capable of giving free, informed and express consent.

Exclusion Criteria:

* Patient with another associated ophthalmological disease, apart from a simple cataract already operated on or operated simultaneously with NDPS or the Xen® break without complications during or after the operation
* History of filtering surgery, history of vitrectomy
* Closed-angle glaucoma
* Pseudo capsular exfoliation (connective tissue disease affecting the eye)
* Uveitic glaucoma (glaucoma related to inflammation which can itself have an effect on the cornea)
* Prolonged postoperative hypertonia (7 days)> 40 mmHG (because this can damage the cells of the cornea)
* Pre-existing endothelial dystrophy, irido-corneo-endothelial syndrome (ICE) (glaucoma with corneal pathology)
* Postoperative athalamy (contact between the iris and the cornea generating endothelial cell loss)
* Endothelial cell count <1000 cells
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
To assess the impact of the type of intervention (NPDS or XEN® placement) on endothelial cell loss 2 years after the intervention | 2 years
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density

SECONDARY OUTCOMES:
Evaluate the impact of the type of intervention on endothelial cell loss after surgery procedure | 1 year postoperative
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density
Evaluate the impact of the type of intervention on endothelial cell loss after surgery procedure | 2 years postoperative
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density
Evaluate the impact of the type of intervention on endothelial cell loss after surgery procedure | 3 years postoperative
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density
Evaluate the impact of the type of intervention on endothelial cell loss after surgery procedure | 4 years postoperative
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density
Evaluate the impact of the type of intervention on endothelial cell loss after surgery procedure | 5 years postoperative
  Difference between the two eye groups in terms of loss of endothelial cell density calculated relative to basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 10% after surgery procedure | 2 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 10% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 10% after surgery procedure | 3 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 10% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 10% after surgery procedure | 4 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 10% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 10% after surgery procedure | 5 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 10% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 20% after surgery procedure | 2 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 20% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 20% after surgery procedure | 3 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 20% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 20% after surgery procedure | 4 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 20% calculated from basal cell density
Evaluate the impact of the type of intervention on the incidence of cell loss of more than 20% after surgery procedure | 5 years postoperative
  Difference between the two eye groups in terms of percentage cell loss ≥ 20% calculated from basal cell density
Evaluate the impact of the position in the anterior chamber of the XEN implant on cell loss after surgery procedure | 2 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the XEN implant on cell loss after surgery procedure | 3 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the XEN implant on cell loss after surgery procedure | 4 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the XEN implant on cell loss after surgery procedure | 5 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the implant on cell loss after surgery procedure | 1 year postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the implant on cell loss after surgery procedure | 2 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the implant on cell loss after surgery procedure | 3 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the implant on cell loss after surgery procedure | 4 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber
Evaluate the impact of the position in the anterior chamber of the implant on cell loss after surgery procedure | 5 years postoperative
  in the eye group operated with XEN® placement: distribution of cell loss according to the position in the anterior chamber of XEN® determined by OCT photographs of the anterior chamber

CONTACTS AND LOCATIONS:
Overall Officials: Yves LACHKAR, Principal Investigator — Fondation Hôpital Saint-Joseph